CLINICAL TRIAL: NCT05548504
Title: HERAN2 Heterogeneously Hypofractionated Radiotherapy for Locally Advanced NSCLC A Randomised Multicentre Phase II Feasibility Study
Brief Title: Heterogeneously Hypofractionated Radiotherapy for Locally Advanced NSCLC
Acronym: HERAN2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Tine Schytte, Professor, Consultant, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20210172
Record Dates: First submitted 2022-02-14; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer Stage III; Radiotherapy Side Effect; Frailty
Keywords: Locally advanced NSCLC; Radiotherapy; Randomized; Photon><proton therapy; Frailty
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Injuries; Frailty | interventions — Photons; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photon therapy (Active Comparator): 50-66Gy/ 24 fractions, inhomogeneous dose distribution Photon therapy
  Interventions: Radiation: Photon
- Proton therapy (Experimental): 50-66Gy/ 24 fractions, inhomogeneous dose distribution Proton therapy
  Interventions: Radiation: Proton

INTERVENTIONS:
Radiation: Photon — 50-66Gy/ 24 fractions, inhomogeneous dose distribution photon therapy
  Arms: Photon therapy
Radiation: Proton — 50-66Gy/ 24 fractions, inhomogeneous dose distribution proton therapy
  Arms: Proton therapy

SUMMARY:
Aim To test if proton therapy can improve survival compared to photon therapy in patients with locally advanced NSCLC who are not candidates for standard definitive chemo-radiotherapy.

Hypothesis The trial hypothesis is that proton therapy is less toxic than photon therapy in fragile patients and that this difference will mitigate to a difference in overall survival.

Design Multicentre, randomized phase II study 1:1 Sample size 182 patients (91 in each arm) Treatment Radiotherapy (inhomogeneous dose distribution) 50 Gy/ 24 fraction Endpoint Primary: Overall survival at 12 months Secondary: progression free survival, time to loco-regional and distant failure, pattern of failure, acute and late toxicity, quality of life, patient compliance.

DETAILED DESCRIPTION:
Study aim To evaluate whether a heterogeneous and hypo-fractionated definitive radiotherapy schedule delivered using proton (PT) can improve OS compared to photon (XT) in patients with LA_NSCLC not candidates for standard, long-course chemo-radiotherapy.

Primary endpoint

* OS at 12 months Secondary endpoints
* Progression-free survival
* Time to loco-regional failure
* Time to distant failure
* Pattern of failure
* Acute toxicity
* Late toxicity
* Persistent acute grade 2 or higher lung or esophageal toxicity
* Radiotherapy compliance
* Hospitalization during and up to 6 months after treatment
* Patient reported outcome measures at base-line and during follow-up Exploratory endpoints
* Heart toxicity evaluated by changes in cardiac biomarkers
* Changes in lymphocyte counts

Study design The study is designed as a prospective randomized multicentre phase II study. It includes patients with inoperable locally advanced NSCLC (stage IIB-IIIB) not candidates for standard concomitant chemotherapy. Patients are treated with radiotherapy in 24 fractions, 5 fractions a week. Dose prescription is inhomogeneous with 50 Gy to the clinical target volume (CTV).

Patients will be randomized 1:1 between XT or PT. It will thus be open-label to the patient and the treating physicians.

Systemic therapy Patients can receive induction therapy with platinum doublet. Randomization and stratification Patients will be randomized (1:1) to either XT or PT. Randomization will be performed centrally using an online 24-hour web-based system maintained by the Clinical Trial Office at Odense University Hospital, ensuring allocation concealment to the clinical investigators. Randomization will be stratified for referring centre and histology (squamous cell carcinoma versus other non-squamous cell carcinoma).

Study sample size The study will use a three-outcome design to examine whether use of PT results in improved OS compared to XT. Preliminary data from the HERAN trial indicate that the patient population (patients not candidate for definitive chemo-radiotherapy) will have a 60% survival rate at 12 months following heterogeneously hypo-fractionated XT. We expect that the patients in HERAN will be representative of the patient population in HERAN2, and that survival in the XT arm will be comparative. A 15%-point improvement in 12 months survival (to 75%) is considered clinically relevant in order to definitely take PT forward for this patient group. 174 patients (87 in each arm) will be needed to provide 80% power to demonstrate this difference at 10% (one-sided) significance level, based on simple comparisons of proportions. Due to the fragile patient population at dropout of 5% is expected, and in order to take this into account 182 patients (91 in each arm) will be included.

It is recognized, however, that a smaller difference (corresponding to a lower level of statistical significance) might still be clinically relevant and warrant further examination of PT for this patient group; provided that the treatment is otherwise tolerable for patients (as measured by toxicity, patient uptake, impact on QoL, and post-treatment hospitalizations rate). Hence a phase II three-outcome screening design is used to form the basis of the decision-making process following the completion of the study, based on the work of Hong & Wang (50) and e.g. used in the SYSTEMS-2 trial (51). The proposed sample size will allow for 90% power to detect a 15%-point difference at 20% (one-sided) significance level; or alternatively 80% to detect a 12%-point difference at the same (80%) significance level. A study outcome in favor of PT at the one-sided 20% level - but not the one-sided 10% level - will thus be considered positive only if other study data supports the use of PT.

Study time frame We consider it realistic to enroll 182 patients from all Danish radiotherapy centres in a period of 3 years.

Data management Data will be filed and stored using electronical 'case report forms' (CRFs) in a local database provided by Open Patient Data Explorative Network (OPEN). The informed consent will ensure the investigators/co-investigators access to the patient's electronic records and collect information at baseline and follow-up.

The clinical data will include: date of birth, gender, smoking history, co-morbidity, weight, TNM stage, histology, performance status, status on prescribed drug, as well as baseline blood test. Relevant for handling of the patients. The data will be obtained from patient file and handed over to the researcher.

All dose plans used for patient treatment, including adapted plans, are exported to the national dose plan bank (DCMCollab), from where doses to tumor, lymph nodes and OAR are extracted for analysis.

Baseline PET-CT scans, as well as any CT or PET-CT scans acquired at time of disease recurrence should also be transferred to the dose plan bank.

The data management system ensures compliance with current legislation and regulations on data handling and data safety.

Withdrawal from the study

A patient may be withdrawn from the study if any of the following events occur:

* If, in the opinion of the investigator, withdrawal is necessary for medical reasons
* Major protocol violation according to national GCP guidelines
* Major technical failure according to national GCP guidelines
* Informed consent withdrawal In case of a withdrawal, another patient will be enrolled (with a new patient number). The withdrawn patient will be accounted for in the statistical analysis. The reason for withdrawal should be clearly described, whenever possible and regardless of the reason for withdrawal. Relevant data should be obtained, and all relevant assessments should be completed, preferably according to the schedule for the final assessment. The CRF in REDCap should be completed.

Screening log All centres will keep a screening log of all patients informed about the trial and in case the patient decline to participate, the reason for declining is noted.

Radiotherapy treatment planning is described in detail. Target dose All treatments are delivered in 24 fractions, 5 fractions per week. For the nominal plan, the mean dose to GTV-T and GTV-N should be increased as much as allowed by normal tissue dose constraint but not exceeding a mean dose of 66 Gy in 24 fractions.

Quality assurance is planned in detail for Target and OAR delineation Treatment planning During the trial, dose volume histograms for the included patients will be analyzed yearly (at minimum) via the national dosebank database to avoid systematic discrepancies between centres.

Study procedures and follow-up Evaluations before and during treatment Patients will be evaluated, and treatment toxicity will be registered at baseline and twice during the course of radiotherapy. If the patient has symptoms which need clinical assessment, the patient will get an appointment with a physician.

Baseline registration consists of baseline patient characteristics. Treatment compliance should be recorded at the end of treatment. Patient reported outcome measures will be scored using EORTC C30 and LC13.

Follow-up Patients will be seen every 3rd month during a follow up period of 24 months and thereafter every 6th month until end of study. During the first 24 months, the patient will be examined every 3rd month with a CT-scan and afterwards twice a year. Lung function test will be performed at 3 months and hereafter yearly. An ECG will be performed at baseline as well as at 3 and 12 months. Clinical examinations and evaluation of toxicity will be performed at every occasion. Disease recurrence, site of recurrence, as well as death should be reported; this may be done by local investigators by review of electronic patient records once a year. End of study is 5 years after commencement of radiotherapy.

The follow-up will be performed at local department of oncology.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed LA_NSCLC
* Not candidate for definitive chemo-radiotherapy
* Performance status 0-2
* Signed informed consent
* Able to comply with study and follow-up procedures

Exclusion Criteria:

* Prior radiotherapy to the thorax unless there is no significant overlap of current treatment volumes with previous treatment fields.
* Uncontrolled other malignant disease.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
OS at 12 months after randomization | 12 month after patient randomization
  Overall survival 12 months after randomization

SECONDARY OUTCOMES:
Acute toxicity | 9 months after patient randomization
  Number of patients with acute toxicity, defined as any radiotherapy related toxicity occurring up to 9 months after randomization
Late toxicity | Up to 5 years after patient randomization
  Number of patients with late toxicity, defined as any radiotherapy related toxicity occurring later than 9 months after randomization.
Progression free survival | up to 5 years after patient randomization
  Any progression or recurrence (locoregional or distant) as well as death from any cause, whatever occurs first, will be considered as events
Pattern of faillure | up to 5 years after patient randomization
  First site of failure will be divided in primary tumour, bulky lymph nodes, non-bulky lymph node targets, regional lymph nodes not included in target delineation/ irradiated, and distant failures.
Changes in level of cardiac biomarkers (BNP) | 12 month after patient randomization
  Changes in Brain Natriuretic peptide (BNP),Troponin T (TnT) and I (TnI) from baseline up to 12 months after radiotherapy
Changes in level of cardiac biomarkers (TnI) | 12 month after patient randomization
  Changes in Troponin I (TnI) from baseline up to 12 months after radiotherapy
Changes in level of cardiac biomarkers (TnT) | 12 month after patient randomization
  Changes in Troponin T (TnT) from baseline up to 12 months after radiotherapy
Changes in level of lymphocyte counts | 12 month after patient randomization
  Changes in lymphocyte count before and after RT
Changes in level of ctDNA | within 12 months after patient randomization
  Circulating tumour DNA detection before RT and during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Tine Schytte, PhD, Principal Investigator — Odense University Hospital

IPD SHARING:
Plan to Share IPD: No